CLINICAL TRIAL: NCT00722995
Title: Surgical Treatment for Morbid Obesity by Sleeve Gastrectomy Versus Gastric Bypass. Study Comparing Complications, Efficacy and Quality of Life.
Brief Title: Surgical Treatment for Morbid Obesity by Sleeve Gastrectomy Versus Gastric Bypass
Acronym: SLEEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K060213
Record Dates: First submitted 2008-07-25; First posted 2008-07-28 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Obesity
Keywords: Morbid obesity; Sleeve gastrectomy; Gastric bypass; Complications; Efficacity; Safety; Compare
MeSH Terms: conditions — Obesity; Obesity, Morbid | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Sleeve gastrectomy
  Interventions: Procedure: Sleeve gastrectomy
- 2 (Active Comparator): Gastric Bypass
  Interventions: Procedure: Gastric Bypass

INTERVENTIONS:
Procedure: Sleeve gastrectomy — Laparoscopic sleeve gastrectomy is a restrictive procedure for the treatment for morbid obesity
  Other Names: SLEEVE
  Arms: 1
Procedure: Gastric Bypass — Laparoscopic gastric bypass is a restrictive and difficult absorption procedure for the treatment of morbid obesity
  Other Names: BYPASS
  Arms: 2

SUMMARY:
The aim of this study is to assess that the sleeve gastrectomy can improve the risk benefit than the gastric bypass

DETAILED DESCRIPTION:
In the obese patient population, the frequency of patients presenting a severe morbid obesity (40 >= BMI <= 50), a super obesity (BMI >50), a super super obesity (BMI>60), and obese patients (BMI>35) with a failure of gastric banding is constantly increasing. In these patients, the surgery risk is proportionate to the weight and / or gastric surgery records.

This risk is high, in bariatric surgery, for gastric bypass procedure. This justifies the evaluation of new procedure to reduce the morbidity allowing the reduction of morbid /mortality associated with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged from 18 to 60 years old
* Patient having given his consent to the use of data from the project
* Patient fulfilling the inclusion criteria for surgery of obesity according to the ANAES (french national health service)
* Patient presenting one of the following criteria:

  * A morbid obesity strict with BMI> 40
  * A super obesity BMI> 50
  * A super super obesity BMI> 60
  * Obese patient in failure following the installation of a gastric banding with BMI> 35
  * obese patient 35>BMI>40 with a comorbidity
* Preliminary agreement during the consultation of a psychiatrist / psychologist

Exclusion Criteria:

* Patient with complications or co morbidities associated involving life to less 6 months
* Patient presenting no anaesthetic indication
* Patient presenting no psychiatric indication for obesity surgery
* Patient not affiliated with a social security scheme
* Pregnant Patient likely to breastfeed in the first year

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 280 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Composite criteria of morbid/mortality | during 18 months and 36 months

SECONDARY OUTCOMES:
Frequency of morbid events | during the follow up
Percentage of excess weight loss | during 18 and 36 months
Frequency of patients having a excess weight loss superior than 50% | during 36 months
Regression of morbidities | during 36 months
Rate serum ghrelin | at inclusion visit, 6, 12, 18 and 36 months
Evaluation of quality of life and scores of precariousness, SF 36, EPWORTH Score, Lequesne' Score, Insecure' Score | at inclusion visit, 6, 12, 18 and 36 months
Frequency of morbid/mortality events | during 36 months
Frequency of patients having excess weight loss superior than 50% | during 18 month

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc CATHELINE, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris / Hôpital De la Fontaine (St Denis)
Locations (1):
- Service de chirurgie digestive / Centre Hospitalier Général de Saint-Denis Delafontaine, Saint-Denis, France